CLINICAL TRIAL: NCT00550602
Title: Tracheobronchomalacia: Treatment Outcomes
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Armin Ernst, MD, BIDMC
Other Study IDs: 2005P000112
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2010-04

CONDITIONS: Tracheomalacia; Tracheobronchomalacia
Keywords: Tracheomalacia; Tracheobronchomalacia; Airway Stabilization; Bronchoscopy; Stent Placement; Tracheobronchoplasty; COPD
MeSH Terms: conditions — Tracheomalacia; Tracheobronchomalacia; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate respiratory symptoms and their impact in the quality of life and after treatment of the respiratory condition (tracheobronchomalacia - TBM).

DETAILED DESCRIPTION:
TBM is an abnormal collapse of the tracheal and bronchial walls. It is characterized by flaccidity of the supporting tracheal and bronchial structures and a significant reduction of airway diameter on expiration seen in the trachea and/or in the mainstem bronchi. Currently there is no available data on the efficacy of central airway stabilization for treating TBM.

Our study would provide this important information and would establish the effect of central airway stabilization on symptoms, functional status, quality of life, lung function and exercise capacity in patients with symptomatic and severe TBM.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of symptomatic tracheal and/or bronchial collapse during bronchoscopy or Dynamic Computed Tomographic study.
* Chronic Obstructive Pulmonary Disease (regardless of severity) and suspicion of tracheal and/or bronchial collapse

Exclusion Criteria:

* inability to follow commands
* Focal extrinsic compression of the trachea/bronchi by mass or other

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population with suspected symptomatic tracheal and/or bronchial collapse referred to our institution by a Pulmonologist or Thoracic Surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2002-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of central airway stabilization on symptoms and quality of life in patients with symptomatic and severe tracheobronchomalacia. | At 10-14 days post-stent ; at 3 months and yearly post-tracheobronchoplasty

SECONDARY OUTCOMES:
To evaluate the effect of central airway stabilization on lung function, exercise capacity and functional status. | At 10-14 days post-stent ; at 3 months and yearly post-tracheobronchoplasty

CONTACTS AND LOCATIONS:
Overall Officials: Armin Ernst, M.D. FCCP, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center- Division of Interventional Pulmonology, Boston, Massachusetts, United States

REFERENCES:
- [Result] Ernst A, Majid A, Feller-Kopman D, Guerrero J, Boiselle P, Loring SH, O'Donnell C, Decamp M, Herth FJ, Gangadharan S, Ashiku S. Airway stabilization with silicone stents for treating adult tracheobronchomalacia: a prospective observational study. Chest. 2007 Aug;132(2):609-16. doi: 10.1378/chest.06-2708. PMID 17699133
- [Derived] Ernst A, Odell DD, Michaud G, Majid A, Herth FFJ, Gangadharan SP. Central airway stabilization for tracheobronchomalacia improves quality of life in patients with COPD. Chest. 2011 Nov;140(5):1162-1168. doi: 10.1378/chest.10-3051. Epub 2011 Aug 25. PMID 21868463
- [Derived] Odell DD, Shah A, Gangadharan SP, Majid A, Michaud G, Herth F, Ernst A. Airway stenting and tracheobronchoplasty improve respiratory symptoms in Mounier-Kuhn syndrome. Chest. 2011 Oct;140(4):867-873. doi: 10.1378/chest.10-2010. Epub 2011 Apr 14. PMID 21493699
- [Derived] Majid A, Guerrero J, Gangadharan S, Feller-Kopman D, Boiselle P, DeCamp M, Ashiku S, Michaud G, Herth F, Ernst A. Tracheobronchoplasty for severe tracheobronchomalacia: a prospective outcome analysis. Chest. 2008 Oct;134(4):801-807. doi: 10.1378/chest.08-0728. PMID 18842912